CLINICAL TRIAL: NCT04662957
Title: The Effectiveness of Multi Strain Probiotic Preparation in Patients With Diarrhea Predominant Irritable Bowel Syndrome - Randomized Double Blide Placebo Controlled Study
Brief Title: Multi Strain Probiotic Preparation in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Memorial Health Institute, Poland (Other)
Collaborators: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Bożena Cukrowska, Prof. MD, PhD, Children's Memorial Health Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MBX02/2019/P
Record Dates: First submitted 2020-12-09; First posted 2020-12-10 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Irritable Bowel Syndrome With Diarrhea; Effects of Probiotics
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic preparation (Experimental): Multi-strain probiotic mixture. The daily dose was five billion (2 capsules/day).
  Interventions: Dietary Supplement: Multi-strain probiotic mixture of four Bifidobacterium, five Lactobacillus and one Streptococcus species or placebo
- Maltodextrin (Placebo Comparator): Maltodextrin comparable in color, texture and taste to the probiotic mixture (2 capsules/day).
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Multi-strain probiotic mixture of four Bifidobacterium, five Lactobacillus and one Streptococcus species or placebo — Oral supplementation with multi-strain probiotic preparation
  Arms: Probiotic preparation
Dietary Supplement: Maltodextrin — Maltodextrin as placebo
  Arms: Maltodextrin

SUMMARY:
Irritable bowel syndrome (IBS) is one of the most common functional gastrointestinal disorders characterized by recurrent abdominal pain associated with defecation or a change in bowel habits without any structural abnormalities. Despite extensive research, the pathogenesis of IBS has not been clearly elucidated yet. Recent studies have shown that disturbed gut microbiota may promote the development and maintenance of IBS. Significant changes in the microbial communities of healthy controls vs IBS patients have been reported in several studies. These findings promoted the research on probiotics for the treatment of IBS. Probiotics are live microorganisms which, when administered at the right dose, have a positive effect on human health. The currently published systemic reviews and meta-analyses of randomized clinical trials have indicated that probiotics have beneficial clinical effects and can help to reduce global and specific IBS symptoms significantly. However, the effect depends on the specific composition of the probiotic preparation, and some meta-analyzes indicate that multi-strain preparations are more effective than single-strain preparations. Therefore, further research is highly anticipated. The purpose of the current clinical trial is to assess the effectiveness of multi-strain probiotic preparation in patients with diarrhea predominant IBS (IBS-D).

ELIGIBILITY:
Inclusion Criteria:

* diarrhea-predominant irritable bowel syndrome (IBS-D)
* at least moderate form of IBS-D assessed using IBS-SSS, i.e. with score >175
* male and female subjects of Caucasian race
* age between 16 and 70 years (inclusive)
* good physical, medical and mental status estimated on the basis of the medical history and a general clinical examination
* results of laboratory tests (hematology, clinical chemistry, serology, and urinalysis) within the normal range of the local laboratory or considered non-clinically significant by the investigator
* patients who have provided freely their own written informed consent
* patients available for the whole study period
* patients who are able to follow strictly the instructions of the investigational team regarding the study procedures and to fulfil the requirements of the protocol
* the following medications are permitted during the course of the study, as long as they are used at a constant dosage and are commenced at least 1 month prior to study start: birth control pill, or depot intramuscular contraceptive preparation, estrogen-progesterone replacement therapy, L-thyroxine, low-dose antidepressants (up to 25 mg day of amitriptyline, nortriptyline, or selective serotonin reuptake inhibitor), low-dose antihypertensives in the diuretic, angiotensin-converting enzyme inhibitor or angiotensin II inhibitor classes
* patients are allowed to take spasmolytic drugs on an ad hoc basis

Exclusion Criteria:

* other than IBD-D types of IBD
* mild type of IBS-D (<175 points in IBS-SSS scale)
* the use of probiotics within last three months
* the treatment with antibiotics within last three months
* a concurrent severe illness (malignancies, uncontrolled hypertension and diabetes mellitus, hepatic, renal or cardiac dysfunctions, serious neurological disorders, psychosis, respiratory disorders such as asthma, chronic obstructive pulmonary disease, hyper- or hypothyroidism)
* chronic bowel disorders other than IBS, including inflammatory bowel diseases, gastroenteritis, stomach and duodenal ulcers, celiac diseases;
* pregnancy or lactation
* diagnosed lactose intolerance
* the use of motility drugs or dietary fiber supplements within 2 weeks before study start
* plan to have surgery during the time of the study
* a history of alcohol or drug abuse
* taking anti-coagulant medications
* participation in another clinical trial within last three months
* patients who will receive antibiotics during the study

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in severity of IBS symptoms using IBS Severity Scoring System (IBS-SSS) | From baseline at 4 and 8 weeks of intervention
  IBS-Severity Scoring System is a 5-question survey that asks: 1. the severity of abdominal pain, 2. frequency of abdominal pain, 3. severity of abdominal distention, 4.dissatisfaction with bowel habit, and 5. interference with quality of life over the past 10 days. Subjects respond to each question on a 100-point visual analogue scale. Each of the five question generates a maximum score of 100 point, and total scores can range from 0-500 with higher scores indicating severe symptoms. A decrease of 30 points is associated with a clinically meaningful improvement.
Improvement or worsening of IBS global symptoms using Global Improvement Scale (IBS-GIS) | From baseline at 4 and 8 weeks of intervention
  IBS-Global Improvement Scale asseses IBS symptoms using a patient-defined 7 point Linkert scale ranging from symptoms substantially worse to substantially improved.
  Patients answer the question "Have you felt any change in the severity of your symptoms over the past 7 days compared to how you felt before the medicine was given?
  The answers are recorded based on the 7-point scale:
  1. I feel that the symptoms have worsened significantly
  2. I feel that the symptoms have moderately worsened
  3. I feel that the symptoms have slightly worsened
  4. I feel no change
  5. I feel a slight improvement
  6. I feel moderate improvement
  7. I feel significant improvement
  IBS-GIS score indicates: improvement if is >4 or worsening if is<4, no change if is 4
Changes in adequate relief of IBS symptoms (IBS-AR) | From baseline at 4 and 8 weeks of intervention
  IBS-Adequate Relief (IBS-AR) is a dichotomous single item that asks participants "Over the past week (7 days) have you had adequate relief of your IBS symptoms? The answer is YES or NO.

SECONDARY OUTCOMES:
Changes in type of stools | From baseline for 8 weeks of intervention
  ype of stool assessed before intervention and then 3 times a week. Type of stools assessed using the Bristol Stool Scale. Bristol Scale is designed to classify faeces into seven groups: type 1-2 indicate constipation, type 3-4 are "normal" stools; type 5-7 indicate diarrhea.
Changes in number of bowel movements per day | From baseline for 8 weeks of intervention
  Number of bowel movements per day assessed before intervention and then 3 times a week
Changes in severity of pain | From baseline for 8 weeks of intervention
  The severity of pain assessed before intervention and then 3 times a week using a patient-defined 5 point Linkert scale: point 0 - no pain, and 1-4 the severity of pain with higher scores indicating worse pain
Changes in flatulence | From baseline for 8 weeks of intervention
  The severity of flatulence assessed before intervention and then 3 times a week using a patient-defined 5 point Linkert scale: point 0 - no flatulence, and points1-4 with higher scores indicating worse flatulence
Changes in feeling of incomplete evacuation of stool | From baseline for 8 weeks of intervention
  The severity of incomplete evacuation of stool assessed before intervention and then 3 times a week using a patient-defined 5 point Linkert scale: point 0 - no feeling of incomplete evacuation of stool, and points1-4 with higher scores indicating worse feeling of incomplete evacuation of stool
Changes in the occurrence of adverse events | From baseline for 8 weeks of intervention
  The number and the type of adverse events assessed before intervention and then 3 times a weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Memorial Health Institute, Warsaw, Poland

REFERENCES:
- [Derived] Skrzydlo-Radomanska B, Prozorow-Krol B, Cichoz-Lach H, Majsiak E, Bierla JB, Kanarek E, Sowinska A, Cukrowska B. The Effectiveness and Safety of Multi-Strain Probiotic Preparation in Patients with Diarrhea-Predominant Irritable Bowel Syndrome: A Randomized Controlled Study. Nutrients. 2021 Feb 26;13(3):756. doi: 10.3390/nu13030756. PMID 33652763